CLINICAL TRIAL: NCT00457444
Title: ZU-SkinSIT-001 Single Center Phase I/IIa, Placebo Controlled, Randomized, Double Blind Study to Assess the Clinical Efficacy and Safety of a Novel Method of Specific Allergen Immunotherapy in Grass Pollen Allergic Subjects by Epicutanous Allergen Administration
Brief Title: Study to Assess the Clinical Efficacy and Safety of a Novel Method of Specific Allergen Immunotherapy in Grass Pollen Allergic Subjects by Epicutanous Allergen Administration
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Zurich (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZU-SkinSIT-001
Record Dates: First submitted 2007-04-05; First posted 2007-04-06 (Estimated); Last update posted 2007-04-06 (Estimated); Status verified 2007-04

CONDITIONS: Rhinoconjunctivitis
MeSH Terms: interventions — Propolis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Pollen

SUMMARY:
Primary Objective Comparison of the inhibition of the allergic response assessed by nasal provocation test after epicutanous pollen allergen administration and placebo epicutaneous administration.

Secondary Objectives Comparison of the efficacy of the placebo with that of the epicutanous pollen allergen administration evaluated by visual analog symptom scales (nasal itching, sneezing, rhinorrhea, conjunctival redness, and lacrimation, lung symptoms ), Comparison of the inhibition of the allergic response assessed by skin prick test after epicutanous pollen allergen administration and placebo epicutaneous administration.

* Trial with medicinal product

ELIGIBILITY:
Inclusion criteria:

* Written informed consent
* History of grass pollen allergic rhinitis
* Male and female between 18 years to 65 years
* Positive skin prick test to grass pollen
* Positive nasal provocation test

Exclusion criteria:

* Atopic eczema in history or permanent
* Perennial allergic rhinitis
* Symptoms of infectious disease with rhinitis in between the last 2 weeks
* Surgical intervention in between the last 30 days
* Pregnancy or nursing
* History of HIV or AIDS
* Mastocytosis (cutaneous or systemic)
* Significant cardiovascular disease
* Hypertension (blood pressure > 160 / 95)
* Significant pulmonary, renal and/or hepatic disease
* Significant hematological disorder
* Moderate or severe asthma
* History of malignancy
* History of neurological or psychatric disease
* Autoimmune disease
* Antihistamines with longed half-lives in the last week
* Systemic or topical steroids for 5 days
* Active infectious disease
* Contraindicated medications: - immunosuppressive agents

  * Betablockers
  * ACE-inhibitors
  * Tricyclic antidepressants
  * Daily use of Beta-agonists or steroid inhalers
* Participation in another clinical trial /study in between the last 60 days
* Participation in another clinical trial / study at the moment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35
Dates: Start 2005-12; Study Completion 2006-11

PRIMARY OUTCOMES:
efficacy

CONTACTS AND LOCATIONS:
Overall Officials: Studienregister MasterAdmins, Study Director — UniversitaetsSpital Zuerich
Locations (1):
- University Hospital Zurich, Zurich, Switzerland